CLINICAL TRIAL: NCT05362006
Title: The Effects of a TENS System (Transcutaneous Electric Nerve Stimulation) on Spasticity and Muscular Oxygenation in Patients With Multiple Sclerosis (ENNOX Study)
Brief Title: Exopulse Mollii Suit, Spasticity & Tissue Oxygenation
Acronym: ENNOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-A01665-36
Record Dates: First submitted 2022-01-24; First posted 2022-05-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Oxygenation; Muscles; Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds.
  Interventions: Device: Exopulse Mollii Suit
- Sham (Sham Comparator): In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Interventions: Device: Exopulse Mollii suit (sham)

INTERVENTIONS:
Device: Exopulse Mollii Suit — Exopulse Mollii suit is a new assistive device that has been developed by Exoneural Network (initially Inerventions AB), a Swedish med-tech company. Exopulse Mollii suit is a full-body garment with integrated 58 electrodes that can transcutaneously stimulate 40 groups of muscles.
  This stimulation is not intended to obtain a motor effect (contraction of the muscles in question), but rather to decrease the spasticity in spastic muscles by activating the antagonistic muscles via the physiological mechanism of reciprocal inhibition. The device is CE labelled and is intended to use for reducing spasticity and improving blood circulation. The outfit is very easy to put on, it can be used for one hour every day and the analgesic effects last 24 hours or more.
  Arms: Active
Device: Exopulse Mollii suit (sham) — In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Arms: Sham

SUMMARY:
Spasticity is a frequent and debilitating symptom in patients with multiple sclerosis (MS). Sustained contractile activity, such as that observed in spastic muscles, could reduce the capillary density and induce important changes in the muscular microcirculation, leading to oxidative changes within the muscular tissue. Such changes reflect altered aerobic metabolism and impaired mitochondrial function. The available therapeutic strategies for treating spasticity and related symptoms are usually faced with limited efficacy and numerous side effects. For these reasons, non-invasive stimulation techniques, namely transcutaneous stimulation by means of Exopulse Mollii suit, might be of help in this context.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis according to the 2017 McDonald criteria since at least one month.
* Age between 18 and 75 years.
* Ability to walk freely or with the need of support (expanded disability status scale score (EDSS) < 7.5).
* Being free of relapses in the last three months.
* Being French speaker, able to understand verbal instructions, and affiliated to the national health insurance (sécurité sociale).
* Having spasticity with a score of at least 1+ on the MAS.

Exclusion Criteria:

* Being included in another research protocol during the study period.
* Inability to undergo medical monitor for the study purposes due to geographical or social reasons.
* Having a cardiac stimulator, a ventriculoperitoneal shunt, an intrathecal baclofen pump or other contraindications to using Exopulse Mollii suit.
* Being pregnant
* Having a change in their pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Having a body mass index above 35 Kg/m2
* In case of the introduction of a medical device other than Exopulse Mollii suit during the study period.
* Patients under juridical protection (" mesure de protection judiciare : tutelle, curatelle, sauvegarde de justice ")
* Prisoners.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in oxyhemoglobin level at baseline and at week 2. | This be assessed at baseline, then at week 2.
  Oxygemoglobin level will be evaluated using Near Infrared Technology (NIRS) by means of a PortaMon device. This is a wireless device - PortaMon (Artinis Medical Systems, The Netherlands) that consists of three light emitting diodes, each sending two wavelengths and four channels to measure tissue oxygenation. PortaMon device can assess the level of oxyhemoglobin of the muscle in question.
  All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Changes in deoxyhemoglobin level at baseline and at week 2. | This be assessed at baseline, then at week 2.
  Deoxyhemoglobin level will be evaluated using the same Near Infrared Technology (NIRS) by means of a PortaMon device as previously described. The device can assess the level of deoxyhemoglobin of the muscle in question.
  All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Changes in tissue oxygenation index at baseline and at week 2. | This be assessed at baseline, then at week 2.
  Tissue oxygenation index will be evaluated using NIRS technology. A wireless device PortaMon (Artinis Medical Systems, The Netherlands)- is designed for this purpose, it consists of three light emitting diodes, each sending two wavelengths and four channels to measure tissue oxygenation index.
  All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Change in total hemoglobin level at baseline and at week 2. | This be assessed at baseline and at week 2.
  Total hemoglobin level is the sum of oxyhemoglobin and deoxyhemoglobin. It will be evaluated using Near Infrared Technology (NIRS) by means of a PortaMon device. PortaMon device can assess the level of oxyhemoglobin of the muscle in question. All NIRS measurements will be done while the muscles of interest are kept at complete rest.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | This be assessed at baseline, then at week 2, week 4 and week 8.
  MAS ranges from 0 (normal muscle tone ) to 4 (rigidity)
Numerical Rating Scale of spasticity (NRS) | This be assessed at baseline, then at week 2, week 4 and week 8.
  NRS ranges ranges from 0 (no spasticity) to 10 (worse spasticity that the participant can imagine)
Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) | This be assessed at week 4 and week 8.
  Quality of life will be measured using the 31-item Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL). The MusiQoL questionnaire comprises 31 questions in 9 dimensions (subscales): activities of daily living (ADL, 8 items), psychological well-being (PWB, 4), symptoms (SPT, 4), relationships with friends (RFr, 3), relationships with family (RFa, 3), sentimental and sexual life (SSL, 2), coping (COP, 2), rejection (REJ, 2), and relationships with healthcare system (RHCS, 3). The index score is computed as the mean of these subscale scores. All 9 dimensions and the index score are linearly transformed and standardized on a 0 to 100 scale, where 0 indicates the worst possible level of QoL and 100 indicates the best level.
Changes in oxyhemoglobin level at week 4 and week 8. | This be assessed at week 4 and week 8.
  Oxygemoglobin level will be evaluated using Near Infrared Technology (NIRS) by means of a PortaMon device. This is a wireless device - PortaMon (Artinis Medical Systems, The Netherlands) that consists of three light emitting diodes, each sending two wavelengths and four channels to measure tissue oxygenation. PortaMon device can assess the level of oxyhemoglobin of the muscle in question.
  All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Changes in deoxyhemoglobin level at week 4 and week 8. | This be assessed at week 4 and week 8.
  Deoxyhemoglobin level will be evaluated using the same Near Infrared Technology (NIRS) by means of a PortaMon device as previously described. The device can assess the level of deoxyhemoglobin of the muscle in question.
  All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Changes in tissue oxygenation index at week 4 and week 8. | This be assessed at week 4 and week 8.
  Tissue oxygenation index will be evaluated using NIRS technology. A wireless device PortaMon (Artinis Medical Systems, The Netherlands)- is designed for this purpose, it consists of three light emitting diodes, each sending two wavelengths and four channels to measure tissue oxygenation index.
  All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Changes in total hemoglobin level at week 4 and week 8. | This be assessed at week 4 and week 8.
  Total hemoglobin level is the sum of oxyhemoglobin and deoxyhemoglobin. It will be evaluated using Near Infrared Technology (NIRS) by means of a PortaMon device. PortaMon device can assess the level of oxyhemoglobin of the muscle in question. All NIRS measurements will be done while the muscles of interest are kept at complete rest.
Visual Analog Scale (VAS) pain | This be assessed at baseline, then at week 2, week 4 and week 8.
  VAS ranges ranges from 0 (no pain) to 10 (the worst pain that the participant can imagine)
Mobility will be assessed using the MSWS-12 (Multiple Sclerosis Walking Scale - 12) | This be assessed at week 4 and week 8.
  Subjective changes in walking would be evaluated in patients who can walk by the Multiple Sclerosis Walking Scale - 12 (MSWS-12), a 12-item scale that examines the impact of MS on walking capacity, is a validated patient-reported measure for exploring this outcome.
Mobility will be assessed using the FES-I (Falls Efficacy Scale-International scale) | This be assessed at week 4 and week 8.
  Subjective risk of fall will be assessed in patients who can walk using the French version of the Falls Efficacy Scale-International scale (FES-I) ; a 14-item scale that assesses the perceived risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No